CLINICAL TRIAL: NCT05328765
Title: ACTION HIV (Anal Cancer TherapIes and Outcomes iNitiative for Patients Living With and Without HIV): A Global Record of Patients With Anal Squamous Cell Carcinoma With and Without HIV Infection
Brief Title: A Global Record of Patients With Anal Squamous Cell Carcinoma With and Without HIV Infection
Acronym: ACTION HIV
Status: Recruiting | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: LACOG 0421
Record Dates: First submitted 2022-04-05; First posted 2022-04-14 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-07

CONDITIONS: Anal Squamous Cell Carcinoma; HIV Infections
Keywords: HIV Infections; Anal Squamous Cell Carcinoma
MeSH Terms: conditions — Anus Neoplasms; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — We will also note whether tumor tissue is available from pre-treatment biopsy at the participating center to plan future translational studies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With HIV Infection: Patients with CCA with HIV infection,
- Without HIV Infection: Patients with CCA without HIV infection,

SUMMARY:
Due to the scarcity of data on prognostic and predictive influence on CCA, epidemiological studies evaluating these factors need to be developed in patients with CCA. Therefore, the investigators want to evaluate the profile of patients in the real world and from various parts of the world, describing prognostic factors such as CD4 dosage, time of HIV infection, evaluation of viral load, diagnosis of AIDS, geographic region of diagnosis and treatment, clinical staging, medications concomitant with QRT (risk of drug interactions), comorbidities (possible impact on dose-intensity), use of HAART, time of use of HAART, radiotherapy modality (conventional 3D vs Modulated Beam Intensity [IMRT], response to Nigro vs CTII regimens, as well as comparing clinical outcomes with patients without HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Confirmed histological diagnosis of anal canal squamous cell carcinoma. Basaloid subtype is accepted
* Have underundered serological test for HIV infection
* Any clinical stage

Exclusion Criteria:

* Lack of data on treatments and clinical outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentially eligible patients will be screened through the administrative lists of participating centres. Based on convenience and viability, we estimate to accumulate 300 patients with CCA with and without HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Median disease-free survival | 3 years
  Defined as time from Day 1 from initiation of treatment (or definition of exclusive supportive care) to tumor death or recurrence. Disease-free survival at 3 years after initiation of treatment: proportion of patients free of local or metastatic disease at 3 years after treatment termination according to imaging tests (chest, abdomen and pelvis scans) and clinical examination of anal inspection
Complete clinical response | 6 months
  Absence of neoplasia on magnetic resonance imaging (preferred) or computed tomography of the pelvis and on clinical examination of anal inspection 6 months after the end of QRT or RT isolated
Overall survival | From first date of treatment to date of death from any cause, assessed up to 3 years.
  Defined as the date from the D1 of treatment (or exclusive supportive care) to death from any cause; living patients at the time of the analysis will be censored.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Riechelmann, Principal Investigator — Brazilian Group of Gastrointestinal Tumors
Locations (1):
- A.C. Camargo Cancer Center, São Paulo, Brazil